CLINICAL TRIAL: NCT02541968
Title: Internet-based vs Face-to-face Cognitive Behavioural Therapy for Obsessive-compulsive Disorder - a Randomized Controlled Non-inferiority Trial
Brief Title: Internet-based vs Face-to-face Cognitive Behavioural Therapy for Obsessive-compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Rück, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OCD F2F vs ICBT
Record Dates: First submitted 2015-08-24; First posted 2015-09-04 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Obsessive-compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Face-to-face CBT (Active Comparator): 16 sessions of individual CBT delivered in 14 weeks.
  Interventions: Behavioral: Cognitive-behavioral therapy (face-to-face)
- Internet-based CBT (Experimental): Internet-based CBT (ICBT) with therapist support (14 weeks).
  Interventions: Behavioral: Internet-based Cognitive-behavioral therapy
- ICBT without therapist support (Experimental): Internet-based CBT without therapist support (14 weeks).
  Interventions: Behavioral: Internet-based Cognitive-behavioral therapy without therapist support

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy (face-to-face)
  Other Names: CBT
  Arms: Face-to-face CBT
Behavioral: Internet-based Cognitive-behavioral therapy — With therapist support
  Other Names: ICBT
  Arms: Internet-based CBT
Behavioral: Internet-based Cognitive-behavioral therapy without therapist support
  Arms: ICBT without therapist support

SUMMARY:
Randomized controlled non-inferiority trial comparing therapist-guided Internet-based Cognitive behavioral therapy (ICBT), self-guided ICBT, and individual face-to-face (f2f) CBT for Obsessive-Compulsive Disorder (OCD) in adults.

The primary objective is to evaluate whether ICBT is a non-inferior treatment option compared to the best possible available treatment for OCD, individual face to face (f2f) CBT. A second objective is to compare the efficacy of self-guided vs. therapist-guided ICBT. As this question has cost implications for the health system, a third objective is to carry out a health economic evaluation of both forms of ICBT, in relation to the gold standard f2f CBT. A fourth objective is to explore whether ICBT is equally suited for clinic-referred cases compared to self-referred patients. Finally, a fifth objective is to investigate whether genetic markers, in combination with clinical variables, can be employed to predict treatment outcomes with CBT in general.

Research Questions:

Q1: Is therapist-guided internet-based CBT (ICBT) for OCD non-inferior to face-to-face (f2f) CBT with regard to OCD symptoms, function and quality of life?

Q2: Is entirely self-guided ICBT non-inferior to f2f CBT with regard to OCD symptoms, function and quality of life?

Q3: Is ICBT a cost-effective treatment, compared to f2f CBT?

Q4: Is there a difference in treatment outcome between self-referred and clinical referred patients?

Q5: Can clinical variables and genetic markers be useful to predict which patients will benefit from CBT?

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age,
* Internet access,
* primary diagnosis of OCD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5),
* Written consent of participation in the study.

Exclusion Criteria:

* Other psychological treatment for OCD during the treatment period,
* Adjustment of concurrent psychotropic medication within the last two months,
* bipolar disorder,
* psychosis,
* alcohol or substance dependence,
* completed CBT for OCD in the last 12 months,
* hoarding disorder or OCD with primary hoarding symptoms,
* suicidal ideation,
* subjects that lack the ability to read written Swedish or lack the cognitive ability to assimilate to the written material,
* Autism spectrum disorder,
* organic brain disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09-03 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | Change from baseline to treatmentweek 2, 4, 6, 8, 10 , 12, 15 and 3- and 12-month follow-up.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
Global Assessment of Functioning (GAF) | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
Structured Clinical Interview for DSM-5 (SCID-5) obsessive-compulsive and related disorders Structured Clinical Interview for DSM-5 (SCID-5) obsessive-compulsive and related disorders | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
  Diagnostic status
Yale-Brown Obsessive-Compulsive Scale - self-rated (Y-BOCS) | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
Obsessive-Compulsive Inventory - Revised (OCI-R) | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
Sheehan Disability Scale (SDS) | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
Montgomery-Åsberg Depression Rating Scale - self-rated (MADRS-S) | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
Euroqol (EQ-5D) | Change from baseline to treatmentweek 15, 3- and 12-month follow-up.
Clinical Global Impression - Improvement (CGI-I) | Treatmentweek 15, 3- and 12-month follow-up.
Insomnia Severity Index (ISI) | Treatmentweek 15, 3- and 12-month follow-up.
Treatment credibility scale | Change from baseline to treatmentweek 2.
Satisfaction with treatment scale | Treatmentweek 15
TiC-P | Treatmentweek 0, 15, 3- and 12-month follow-up.
  Self-rated questionnaire on healthcare utilization and productivity losses in patients with a psychiatric disorder
Safety Monitoring Uniform Report Form (SMURF) | Treatmentweek 2, 4, 6, 8, 10 , 12, 15 and 3- and 12-month follow-up.
Patient EX/RP Adherence Scale (PEAS) | Treatmentweek 6 and 15
Working Alliance Inventory - short revised | Change from baseline to treatment week 6 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rück, Principal Investigator — Karolinska Institutet
Locations (1):
- Mottagningen för Tvångssyndrom, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson E, Hedman E, Enander J, Radu Djurfeldt D, Ljotsson B, Cervenka S, Isung J, Svanborg C, Mataix-Cols D, Kaldo V, Andersson G, Lindefors N, Ruck C. D-Cycloserine vs Placebo as Adjunct to Cognitive Behavioral Therapy for Obsessive-Compulsive Disorder and Interaction With Antidepressants: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Jul;72(7):659-67. doi: 10.1001/jamapsychiatry.2015.0546. PMID 25970252
- [Background] Andersson E, Steneby S, Karlsson K, Ljotsson B, Hedman E, Enander J, Kaldo V, Andersson G, Lindefors N, Ruck C. Long-term efficacy of Internet-based cognitive behavior therapy for obsessive-compulsive disorder with or without booster: a randomized controlled trial. Psychol Med. 2014 Oct;44(13):2877-87. doi: 10.1017/S0033291714000543. Epub 2014 Mar 14. PMID 25066102
- [Result] Lundstrom L, Flygare O, Andersson E, Enander J, Bottai M, Ivanov VZ, Boberg J, Pascal D, Mataix-Cols D, Ruck C. Effect of Internet-Based vs Face-to-Face Cognitive Behavioral Therapy for Adults With Obsessive-Compulsive Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e221967. doi: 10.1001/jamanetworkopen.2022.1967. PMID 35285923
- [Derived] Ruck C, Lundstrom L, Flygare O, Enander J, Bottai M, Mataix-Cols D, Andersson E. Study protocol for a single-blind, randomised controlled, non-inferiority trial of internet-based versus face-to-face cognitive behaviour therapy for obsessive-compulsive disorder. BMJ Open. 2018 Sep 5;8(9):e022254. doi: 10.1136/bmjopen-2018-022254. PMID 30185575